CLINICAL TRIAL: NCT04510324
Title: Plant-Based Meat vs Animal "Red" Meat: a Randomized Cross-over Trial
Brief Title: Plant-Based Meat vs Animal "Red" Meat Trial
Acronym: FOOD-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: João Pedro Ferreira, MD (Unknown)
Responsible Party: Principal Investigator, Abhinav Sharma, Cardiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-6374
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Response
Keywords: TMAO; Red meat; Plant-base nutrition; Cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, single-blinded cross-over trial including healthy adult participants (N=40, omnivores, aged between 25 and 65 years, and with a body mass index (BMI) between 20 and 40 kg/m2 (see participation criteria below). Following one week of a meat, egg, and seafood free diet ('washout'), participants will be randomized to either red meat (cow burger) or plant meat (plant-based burger) for one week. Following this, participants will under go another week of diet washout and will then be crossed over to the other meat burger for one week. The primary outcome will be the within-group change in the TMAO levels.
Who Masked: Participant
Masking Description: Patients will be randomized in a 1:1 ratio. Randomization will be performed within the electronic database system at the time of enrollment using a random number generator, an approach we have used successfully in other clinical trials. The participants will be blinded to the intervention assignment (single blinded study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red meat patties (Active Comparator): Participants will be randomized to group 1: Red meat, ''Costco Kirkland Signature 1/4 lb Ground Beef Patties'' (Beef burger). Participants will be given two patties per day.
  Interventions: Other: Red meat patties group
- Plant-based patties (Experimental): Participants will be randomized to group 2: plant-based burger which contains no animal products. The Plant-based burger selected is ''Beyond Burger" (https://www.beyondmeat.com/products/the-beyond-burger/ ). Participants will be given two patties per day.
  Interventions: Other: Plant-based patties group

INTERVENTIONS:
Other: Red meat patties group — 1. Baseline Visit: day -7 before randomization
  * Clinical history
  * Refrain from seafood, eggs, fish or meat, for 7-day ("washout") prior to Day 1. 2. Day 1 Randomization
  * Randomization to 1 of 2 interventions: plant-based or meat burgers
  * 6 days-worth of burgers will be delivered to the participant's house 3. Day 1-6:
  * The participant will be asked to eat a specific randomized diet for 6 days 5. Days 7
  * Physical exam (weight, BP, HR)
  * Food questionnaire
  * Blood draw: Circulating TMAO, Total, LDL, and HDL cholesterol, Creatinine, High-sensitivity c-reactive protein
  * Urine Collection - TMAO 6. Day 7-14: Washout 7. Day 14: Patties delivery 8. Day 14-20: Assigned diet for 6 days 9. Days 20: Same as day 7
  Arms: Red meat patties
Other: Plant-based patties group — Same as above
  Arms: Plant-based patties

SUMMARY:
To assess the changes in the circulating levels of TMAO after 1-week of beef or plant-based burger diet.

DETAILED DESCRIPTION:
Single-center, randomized, single-blinded cross-over trial including healthy adult participants (N=40, omnivores, aged between 25 and 65 years, and with a body mass index (BMI) between 20 and 40 kg/m2 (see participation criteria below). Participants will be randomized to either red meat (cow burger) or plant "meat" (plant-based burger). The primary outcome will be the within-group change in the TMAO levels.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 25 years and ≤65 of age
* BMI ≥20 Kg/m2 and ≤40 Kg/m2
* No known kidney disease
* No antibiotics in the previous 30 days

Exclusion Criteria:

* Any person who does not meet the above criteria and/or who refuses to participate
* Food allergies (specific ingredients contained in the patties)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in TMAO levels | Baseline Day 6-7-20-21
  Blood and urine analysis will be performed to determine TMAO levels after each intervention

SECONDARY OUTCOMES:
Change in total, LDL, and HDL cholesterol | Baseline Day 6-7-20-21
  Blood and urine analysis will be performed to determine cholesterol levels after each intervention
Change in high-sensitivity c-reactive protein | Baseline Day 6-7-20-21
  Blood and urine analysis will be performed to determine c-reactive protein levels after each intervention
Change in systolic and diastolic blood pressure | Baseline Day 6-7-20-21
  Assessment of blood pressure
Change in heart rate | Baseline Day 6-7-20-21
  Assessment of heart rate

OTHER OUTCOMES:
Adherence of diet | Baseline Day 6-7-20-21
  Self-reported completion of dietary intervention
Tolerance of diet | Baseline Day 6-7-20-21
  Self-reported tolerance of dietary intervention
Identification of study intervention | Baseline Day 6-7-20-21
  Self-reported identification of dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sharma, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The coded data will be securely shared with Dr. João Pedro Ferreira at the University of Lorraine, Clinical Research Center of Nancy in France.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Undetermined

REFERENCES:
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Schiattarella GG, Sannino A, Toscano E, Giugliano G, Gargiulo G, Franzone A, Trimarco B, Esposito G, Perrino C. Gut microbe-generated metabolite trimethylamine-N-oxide as cardiovascular risk biomarker: a systematic review and dose-response meta-analysis. Eur Heart J. 2017 Oct 14;38(39):2948-2956. doi: 10.1093/eurheartj/ehx342. PMID 29020409
- [Background] Bennett BJ, de Aguiar Vallim TQ, Wang Z, Shih DM, Meng Y, Gregory J, Allayee H, Lee R, Graham M, Crooke R, Edwards PA, Hazen SL, Lusis AJ. Trimethylamine-N-oxide, a metabolite associated with atherosclerosis, exhibits complex genetic and dietary regulation. Cell Metab. 2013 Jan 8;17(1):49-60. doi: 10.1016/j.cmet.2012.12.011. PMID 23312283
- [Background] Warrier M, Shih DM, Burrows AC, Ferguson D, Gromovsky AD, Brown AL, Marshall S, McDaniel A, Schugar RC, Wang Z, Sacks J, Rong X, Vallim TA, Chou J, Ivanova PT, Myers DS, Brown HA, Lee RG, Crooke RM, Graham MJ, Liu X, Parini P, Tontonoz P, Lusis AJ, Hazen SL, Temel RE, Brown JM. The TMAO-Generating Enzyme Flavin Monooxygenase 3 Is a Central Regulator of Cholesterol Balance. Cell Rep. 2015 Jan 20;10(3):326-338. doi: 10.1016/j.celrep.2014.12.036. Epub 2015 Jan 15. PMID 25600868
- [Background] Wang Z, Roberts AB, Buffa JA, Levison BS, Zhu W, Org E, Gu X, Huang Y, Zamanian-Daryoush M, Culley MK, DiDonato AJ, Fu X, Hazen JE, Krajcik D, DiDonato JA, Lusis AJ, Hazen SL. Non-lethal Inhibition of Gut Microbial Trimethylamine Production for the Treatment of Atherosclerosis. Cell. 2015 Dec 17;163(7):1585-95. doi: 10.1016/j.cell.2015.11.055. PMID 26687352
- [Background] Roberts AB, Gu X, Buffa JA, Hurd AG, Wang Z, Zhu W, Gupta N, Skye SM, Cody DB, Levison BS, Barrington WT, Russell MW, Reed JM, Duzan A, Lang JM, Fu X, Li L, Myers AJ, Rachakonda S, DiDonato JA, Brown JM, Gogonea V, Lusis AJ, Garcia-Garcia JC, Hazen SL. Development of a gut microbe-targeted nonlethal therapeutic to inhibit thrombosis potential. Nat Med. 2018 Sep;24(9):1407-1417. doi: 10.1038/s41591-018-0128-1. Epub 2018 Aug 6. PMID 30082863
- [Background] Koeth RA, Wang Z, Levison BS, Buffa JA, Org E, Sheehy BT, Britt EB, Fu X, Wu Y, Li L, Smith JD, DiDonato JA, Chen J, Li H, Wu GD, Lewis JD, Warrier M, Brown JM, Krauss RM, Tang WH, Bushman FD, Lusis AJ, Hazen SL. Intestinal microbiota metabolism of L-carnitine, a nutrient in red meat, promotes atherosclerosis. Nat Med. 2013 May;19(5):576-85. doi: 10.1038/nm.3145. Epub 2013 Apr 7. PMID 23563705
- [Background] Conlon MA, Bird AR. The impact of diet and lifestyle on gut microbiota and human health. Nutrients. 2014 Dec 24;7(1):17-44. doi: 10.3390/nu7010017. PMID 25545101
- [Background] Miller CA, Corbin KD, da Costa KA, Zhang S, Zhao X, Galanko JA, Blevins T, Bennett BJ, O'Connor A, Zeisel SH. Effect of egg ingestion on trimethylamine-N-oxide production in humans: a randomized, controlled, dose-response study. Am J Clin Nutr. 2014 Sep;100(3):778-86. doi: 10.3945/ajcn.114.087692. Epub 2014 Jun 18. PMID 24944063
- [Background] Koeth RA, Lam-Galvez BR, Kirsop J, Wang Z, Levison BS, Gu X, Copeland MF, Bartlett D, Cody DB, Dai HJ, Culley MK, Li XS, Fu X, Wu Y, Li L, DiDonato JA, Tang WHW, Garcia-Garcia JC, Hazen SL. l-Carnitine in omnivorous diets induces an atherogenic gut microbial pathway in humans. J Clin Invest. 2019 Jan 2;129(1):373-387. doi: 10.1172/JCI94601. Epub 2018 Dec 10. PMID 30530985
- [Background] Wang Z, Bergeron N, Levison BS, Li XS, Chiu S, Jia X, Koeth RA, Li L, Wu Y, Tang WHW, Krauss RM, Hazen SL. Impact of chronic dietary red meat, white meat, or non-meat protein on trimethylamine N-oxide metabolism and renal excretion in healthy men and women. Eur Heart J. 2019 Feb 14;40(7):583-594. doi: 10.1093/eurheartj/ehy799. PMID 30535398
- [Background] Mertens E, Markey O, Geleijnse JM, Givens DI, Lovegrove JA. Dietary Patterns in Relation to Cardiovascular Disease Incidence and Risk Markers in a Middle-Aged British Male Population: Data from the Caerphilly Prospective Study. Nutrients. 2017 Jan 18;9(1):75. doi: 10.3390/nu9010075. PMID 28106791
- [Background] Taesuwan S, Cho CE, Malysheva OV, Bender E, King JH, Yan J, Thalacker-Mercer AE, Caudill MA. The metabolic fate of isotopically labeled trimethylamine-N-oxide (TMAO) in humans. J Nutr Biochem. 2017 Jul;45:77-82. doi: 10.1016/j.jnutbio.2017.02.010. Epub 2017 Apr 13. PMID 28433924
- [Background] Janeiro MH, Ramirez MJ, Milagro FI, Martinez JA, Solas M. Implication of Trimethylamine N-Oxide (TMAO) in Disease: Potential Biomarker or New Therapeutic Target. Nutrients. 2018 Oct 1;10(10):1398. doi: 10.3390/nu10101398. PMID 30275434